CLINICAL TRIAL: NCT01519167
Title: Phase IV, Open-Label, Safety Study Evaluating the Use of Dexmedetomidine in Pediatric Subjects Undergoing Procedure-Type Sedation
Brief Title: Open-Label, Safety Study Evaluating the Use of Dexmedetomidine in Pediatric Subjects Undergoing Procedure-Type Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEX-10-16
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2015-08

CONDITIONS: Ultrasound; CT Scans; MRIs
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam; Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — 0.1 - 1.0 mcg/kg/hr IV
Drug: Midazolam — 0.025 - 2 mg/kg IV
Drug: Fentanyl — 0.5 - 3 mcg/kg IV

SUMMARY:
The objective of this study is to evaluate the safety of dexmedetomidine in a pediatric population requiring non-intubated, spontaneous breathing, moderate to deep sedation (NI-MDS) for elective diagnostic or therapeutic procedures, expected to take more than 30 minutes.

DETAILED DESCRIPTION:
This study was designed to evaluate the safety of a continuous infusion of dexmedetomidine (1 mcg/kg loading dose with 0.6 mcg/kg/hr initial maintenance dose and titrated between 0.2-1.0 mcg/kg/hr) administered to subjects requiring non-intubated, spontaneous breathing, moderate to deep sedation (NI-MDS) for elective diagnostic or therapeutic procedures that are expected to take more than 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥28 weeks gestational age and <17 years of age.

   - Preterm subjects ≥28 weeks through <38 weeks, gestational age; (Note: Gestational age will be calculated as the time elapsed between the first day of the last menstrual period to the day of enrollment. If pregnancy was achieved using assisted reproductive technology, gestational age will be calculated by adding 2 weeks to the gestational age as calculated above.)
2. Subject is American Society of Anesthesiologists (ASA) Physical Status I, II or III.
3. Subject requires non-intubated, spontaneous breathing, moderate to deep sedation (NI-MDS) in an operating or procedure room with an an intensivist, anesthesiologist or dental anesthesiologist in attendance.
4. Scheduled for an elective procedure that falls into one of the following three populations:

   * Non-invasive diagnostic/therapeutic procedures (NIDTP): including ultrasound (US), computed tomography (CT) scans, magnetic resonance imaging (MRI), cardiac catheterization, transthoracic echocardiogram (TTE);
   * Minimally invasive diagnostic/therapeutic procedures (MIDTP): including minimally invasive procedures performed under US or CT guidance (e.g. US or CT-guided solid organ biopsy), and routine myocardial biopsies in cardiac transplant recipients;
   * Surgical procedures: including small surgical procedures (e.g. excisions, biopsies) and dental procedures (e.g. extractions, pulpectomy, pediatric rehabilitation dental procedures, filings and crowns).
5. Duration of the procedure is expected to take at least 30 minutes to complete.
6. If female, subject is non-lactating and is either:

   1. Not of childbearing potential, defined as pre-menarche, or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy or hysterectomy.
   2. Of childbearing potential but is not pregnant at time of baseline and is practicing one of the following methods of birth control: oral or parenteral contraceptives, double-barrier method, vasectomized partner, or abstinence from sexual intercourse.
7. Subject's parent(s) or legally acceptable representative(s) has/have voluntarily signed and dated the informed consent document approved by the Institutional Review Board. Assent will be obtained where age-appropriate and according to state regulations.

Exclusion Criteria:

1. Subjects weight at the time of screening is less than 1000 g.
2. Subject has received general anesthesia within 7 days prior to study drug administration.
3. Subject has participated in an experimental/investigational drug study within 30 days prior to study drug administration.
4. Subject has been exposed to dexmedetomidine within 48 hours prior to study drug administration.
5. Subject that has been previously enrolled in this study (DEX-10-16).
6. Subject requires endotracheal intubation or laryngeal mask airway (LMA).
7. Subject is with neurological conditions that in the opinion of the Investigator will preclude reliable assessment of sedation scoring. Examples include, but are not limited to the following: cerebral palsy, autism, severe mental retardation, etc.
8. Subject has central nervous system (CNS) disease with an anticipated potential for increased intracranial pressure, an uncontrolled seizure disorder and/or known psychiatric illness that could confound a normal response to sedative treatment.
9. Subject requires epidural or spinal anesthesia.
10. Subject has received treatment with an alpha-2 agonist or antagonist within 14 days prior to study drug administration.
11. Subject has a known allergy to dexmedetomidine, midazolam or fentanyl.
12. Subject is requiring cardiac catheterization for the purpose of conducting an electrophysiology (EP) evaluation or percutaneous intervention (i.e. angioplasty).
13. Subject for whom opiates, benzodiazepines, dexmedetomidine or other alpha-2 agonists are contraindicated.
14. Subject has received an IV opioid within one hour, or oral/intramuscular (PO/IM) opioid within four hours, prior to the start of study drug administration.
15. Subject has received any pre-induction medication (ie, ketamine, chloral hydrate, benzodiazepines) within 4 hours prior to the start of study drug administration.
16. Subject has acute myocardial infarction recently diagnosed by confirmatory laboratory findings within 6 weeks of screening.
17. Subject has moderate to severe sleep apnea syndrome.
18. Subject has oxygen saturation (SpO2) ≤90% at screening or baseline, except for patients with known cyanotic heart disease undergoing cardiac catheterization.
19. Subject has bradycardia immediately before dosing, according to respective age group.

    * ≥28 weeks to <1 month: Heart Rate (HR) <120 beats per minute (bpm)
    * 1 month to <3 months: HR <100 bpm
    * 3 months to <6 months: HR <90 bpm
    * 6 months to <1 year: HR <80 bpm
    * 1 year to <2 years: HR <70 bpm
    * 2 years to <6 years: HR <60 bpm
    * 6 years to <12 years: HR <55 bpm
    * 12 years to 17 years: HR <50 bpm;

    Note: Subject can be reassessed after 5 minutes
20. Subject has hypotension immediately before dosing, according to respective age group.

    * ≥28 weeks to <1 month: <60 mmHg (systolic blood pressure [SBP])
    * 1 month to <12 months: <70 mmHg (SBP)
    * 1 year to <10 years: <70 + (2 X age in years) mmHg (SBP)
    * 10 years to 17 years: <90 mmHg (SBP);

    Note: Subject can be reassessed after 5 minutes
21. Subject has a presence of second-degree or third-degree heart block at screening or baseline. The presence of a temporary or permanent pacemaker will waive this exclusion criterion.
22. Subject has acute febrile illness, with a temperature (core or tympanic) ≥38.0°C.
23. Subject has any other condition or factor which, in the Investigator's opinion, might increase the risk to the subject.

Ages: 28 Weeks to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Little Rock, Arkansas
  - Anaheim, California
  - Stanford, California
  - Miami, Florida
  - Durham, North Carolina
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Sandy City, Utah
- San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of subjects enrolled was 91, of that 90 subjects received study drug. The remaining 1 subject not treated due to subject being a screen failure.
Groups:
- Dose Level 1: Dexmedetomidine Loading dose 0.1 mcg/kg and Maintenance dose 0.1 mcg/kg/hr
- Dose Level 2: Dexmedetomidine Loading dose 1 mcg/kg and Maintenance dose 0.6 mcg/kg/hr
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2
Started | 1 | 89
Completed | 1 | 81
Not Completed | 0 | 8
Not completed — Diagnostic/TherapeuticProcedureCompleted | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Medical condition changes&deep sedation | 0 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Evaluable Population: All subjects who receive any amount of study drug. All safety analyses will be performed on this population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 1 | 89 | 90
Age, Continuous [Mean (Full Range); unit: years] | 0.1 [0.1 to 0.1] | 7.97 [0.3 to 17.3] | 7.89 [0.1 to 17.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 41 | 41
  Male | 1 | 48 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 23 | 23
  Not Hispanic or Latino | 1 | 66 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 22 | 23
  White | 0 | 60 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Had Success in Sedation
Description: Success in sedation was defined by a combined endpoint which was the combination of the following:
  1. Subject had adequate level of sedation (University of Michigan Sedation Scale [UMSS] score between 1 to 3 [minimally sedated to deeply sedated] or Neonatal Pain, Agitation and Sedation Scale [N-PASS] score between -5 to -2 [Light sedation]) at least 80% of the time the subject was given the study drug.
  2. Subject had successfully completed the procedure without a need for rescue sedation (Midazolam).
  3. Subject had undergone the procedure without artificial ventilation or intervention to restore baseline or normal hemodynamic status
Time Frame: From baseline to end of post-treatment period (approximately 24 hours)
Population: Efficacy Evaluable Population (Participants who received study drug infusion for at least 30 minutes and had no major protocol deviations)
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 1 | 77
participants
  NIDTP (n=1, 40) | 0 | 2
  MIDTP (n=0, 25) | 0 | 0
  Surgical procedures (n=0, 12) | 0 | 0

2. Secondary Outcome: Number of Subjects Not Receiving Rescue Midazolam
Description: Number of subjects who did not receive any rescue midazolam for sedation during the study drug infusion.
Time Frame: During the treatment period, up to approximately 24 hours
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 1 | 77
participants
  NIDTP (n=1, 40) | 1 | 12
  MIDTP (n=0, 25) | 0 | 5
  Surgical procedures (n=0, 12) | 0 | 1

3. Secondary Outcome: Number of Subjects Who Have Undergone Procedures Without Artificial Ventilation or Intervention
Time Frame: During the treatment period, up to approximately 24 hours
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 1 | 77
participants
  NIDTP (n=1, 40) | 1 | 37
  MIDTP (n=0, 25) | 0 | 19
  Surgical procedures (n=0, 12) | 0 | 12

4. Secondary Outcome: Number of Subjects Who Were Adequately Sedated at Least 80% of Time
Description: Subjects who are adequately sedated (UMSS score of 1 to 3 or NPASS score of -5 to -2) at least 80% of the time sedated with the study drug
Time Frame: During the treatment period, up to approximately 24 hours
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 1 | 77
participants
  NIDTP (n=1, 40) | 0 | 21
  MIDTP (n=0, 25) | 0 | 7
  Surgical procedures (n=0, 12) | 0 | 2

5. Secondary Outcome: Time to First Dose of Rescue Midazolam From Start of Dexmedetomidine Infusion
Description: Kaplan-Meier estimates of time in minutes to first dose of rescue midazolam from onset of study drug infusion
Time Frame: During the treatment period, up to approximately 24 hours
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 1 | 77
Hours
  NIDTP (n=1, 40) | NA — There was one subject in this group (n=1) and the subject did not receive rescue midazolam. | 23.5 [16.00 to 28.00]
  MIDTP (n=0, 25) | NA — No subjects were in the MIDTP group | 20.00 [17.00 to 34.00]
  Surgical procedures (n=0, 12) | NA — No subjects were in the surgical procedures group | 20.00 [15.00 to 25.00]

6. Secondary Outcome: Frequency of Midazolam Required for Sedation
Description: Frequency of rescue sedation (midazolam) required to maintain a subject within the target sedation range (UMSS score greater than 1 or N-PASS score less than -2).
Time Frame: During the treatment period, up to approximately 24 hours
Population: Number of subjects who received any amount (mg) of rescue midazolam for sedation in efficacy evaluable population.
Measure: Median (Full Range); unit: Occurrence
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 59
Occurrence
  NIDTP (n=0, 28) |  | 2 [1 to 4]
  MIDTP (n=0, 20) |  | 1 [1 to 2]
  Surgical procedures (n=0, 11) |  | 1 [1 to 2]

7. Secondary Outcome: Frequency of Fentanyl Use for Analgesia
Description: Frequency of rescue analgesia (fentanyl) required from the start of IV sedation to completion of the procedure.
Time Frame: During the treatment period, up to approximately 24 hours
Population: Number of subjects who received any amount (mg) of rescue fentanyl for analgesia in efficacy evaluable population.
Measure: Median (Full Range); unit: Occurrence
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 40
Occurrence
  NIDTP (n=0, 6) |  | 1 [1 to 3]
  MIDTP (n=0, 22) |  | 1 [1 to 5]
  Surgical procedures (n=0, 12) |  | 2.50 [1 to 5]

8. Secondary Outcome: Total Amount of Rescue Sedation (Midazolam)
Description: Total amount of rescue sedation (midazolam) required from the start of IV sedation to completion of the procedure
Time Frame: During the treatment period, up to approximately 24 hours
Population: Number of subjects who received any amount (mg) of rescue midazolam for sedation in efficacy evaluable population.
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 59
milligram
  NIDTP (n=0, 28) |  | 2.62 (1.611)
  MIDTP (n=0, 20) |  | 1.70 (0.767)
  Surgical procedures (n=0, 11) |  | 2.45 (0.907)

9. Secondary Outcome: Total Amount of Rescue Analgesia (Fentanyl)
Description: Total amount of rescue analgesia (fentanyl) required from the start of IV sedation to completion of the procedure
Time Frame: During the treatment period, up to approximately 24 hours
Population: Number of subjects who received any amount (mg) of rescue fentanyl for analgesia in efficacy evaluable population.
Measure: Mean (Standard Deviation); unit: microgram
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 40
microgram
  NIDTP (n=0, 6) |  | 10.83 (8.010)
  MIDTP (n=0, 22) |  | 61.86 (65.740)
  Surgical procedures (n=0, 12) |  | 104.83 (72.007)

10. Secondary Outcome: Number of Subjects Converted to Alternative Sedation or Anesthetic Therapy Due to Failure of Treatment of Study Drug and Rescue Medication
Time Frame: During the treatment period, up to approximately 24 hours
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 1 | 77
Participants
  NIDTP (n=1, 40) | 0 | 0
  MIDTP (n=0, 25) | 0 | 0
  Surgical procedures (n=0, 12) | 0 | 2

ADVERSE EVENTS:
Time Frame: Non-serious adverse events from start of study drug administration until 24(±12) hours following study drug discontinuation. Reported serious adverse events from the time the subject signed informed consent until 30 days after study drug discontinuation.
Arm/Group | Dose Level 1 | Dose Level 2
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/89
Other Adverse Events (participants affected / at risk) | 1/1 | 66/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=1) | Dose Level 2 (N=89)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=1) | Dose Level 2 (N=89)
Bradycardia (Cardiac disorders) | 0 | 4
Tachycardia (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Blood pressure diastolic decreased (Investigations) | 0 | 2
Blood pressure systolic decreased (Investigations) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 3
Somnolence (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 53
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator may not submit the results of the study for publication without the prior written consent of Hospira.